CLINICAL TRIAL: NCT04712617
Title: Sex and Gender Difference in Overlap Syndrome of Functional Gastrointestinal Disorder and the Effect of Genetic Polymorphism in South Korea
Brief Title: Overlap FGIDs and Genetic Polymorphism
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2006-616-128
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Functional Gastrointestinal Disorders; Overlap Syndromes
Keywords: functional gastrointestinal disorder; overlap syndromes; functional dyspepsia; irritable bowel syndrome; non-erosive reflux disease; reflux hypersensitivity
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome; Non-Erosive Reflux Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FGIDs: Patient who were diagnosed with NERD/RH, FD, IBS and their overlaps (NERD/RH-FD, NERD/RH-IBS, FD-IBS, NERD/RH-FD-IBS)
- Healthy controls: Subjects who underwent GI evaluations as part of health check-up or for other problems, such as mild abdominal discomfort or pain for a relatively short period of time, but had no organic problems during GI endoscopy

SUMMARY:
1. To analyze the prevalence of overlap syndromes among NERD or RH, FD, and IBS patients, and to identify and to compare the differences in their characteristics and symptoms, and to determine their risk factors.
2. To identify the differences in clinical features according to sex and gender.
3. To analyze the effect of genetic polymorphisms on overlap FGIDs over long-term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

FGID group

* No organic diseases in routine laboratory tests, abdominal imaging, esophagogastroscopy, and colonoscopy
* NERD or reflux hypersensitivity (RH): typical heartburn occurring at least once a week without visible esophageal mucosal break detected by endoscopy
* FD or IBS: based on the Rome III criteria

Control group

- Subjects who underwent GI evaluations as part of health check-up or for other problems, such as mild abdominal discomfort or pain for a relatively short period of time, but had no organic problems during GI endoscopy

Exclusion Criteria:

* history of GI surgery except appendectomy
* inflammatory bowel disease
* any malignancy, or systemic diseases requiring chronic medication except for hypertension and diabetes mellitus
* pregnant or lactating women
* hepatic, biliary, or psychiatric disorders requiring medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient who were diagnosed with NERD/RH, FD, IBS and their overlaps (NERD/RH-FD, NERD/RH-IBS, FD-IBS, NERD/RH-FD-IBS) and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Symptom severity score (5 Likert scale, from 0 to 4) | per 16 years
  FGID symptom severity score score by K-BDQ
Hospital anxiety and depression scale (HADS) | per 16 years
  by HADS questionnaire
Genetic polymorphisms of SLC6A4 5-HTTLPR, GNB3, ADRA2, TNFA, IL10 gene | per 16 years

SECONDARY OUTCOMES:
Prevalence of overlap syndromes among FGIDs(NERD or RH, FD, and IBS) patients | per 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, Professor, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No